CLINICAL TRIAL: NCT06786728
Title: Evaluation of Decongestion Guided By VExUS Score Or Lung Ultrasound For Renal Recovery In Patients With Cardiorenal Syndrome Type-1 : a Randomized Controlled Trial
Brief Title: Decongestion Guided By VExUS Score Or Lung Ultrasound For Renal Recovery In Patients With Cardiorenal Syndrome Type -1
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Asmaa Shahat Mohamedy Behairy, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD8.1.2024
Record Dates: First submitted 2024-12-05; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cardiorenal Syndrome Type 1
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the VEXUS group :in this group we use the vexus score to guide decongestive theapy (Active Comparator): the use of diuretic if vexus score more than 1 at time of enrollement
  Interventions: Drug: frusemide
- the lung US group : we use lung ultrasound score to detect degree of pulmonary congestion (Active Comparator): if lung ultrasound score more than 15 we will start diuretic therapy
  Interventions: Drug: frusemide

INTERVENTIONS:
Drug: frusemide — in this group we use vexus score to asses decongestion in comparison to lung ultrasound in other group

SUMMARY:
the goal of this observational study is to evaluate the role of VEXUS score and lung ultrasound to guide decongestive therapy in patients with cardiorenal syndrome type -1. the main question it aims to answer is: Can the VEXUS score and lung ultrasound guide the efffect of decongestive therapy on KFR and decongestion metrics in patients with CRS-1 compared to standard assesment ?

ELIGIBILITY:
Inclusion Criteria:

* • Patients of both genders aged 18-65 years old.

  * Patients with CRS1 criteria (worsening of renal function due to acute heart failure manifested by : ( Dyspnea , orthopnea ,hypoxia , congested neck veins , oliguria and congestion in imaging.)
  * Patients with Modified lung ultrasound score(LUSS) more than 15.

Exclusion Criteria:

* • Refusal to participate.

  * Patients with renal transplantation.
  * Unknowing baseline creatinine.
  * Patients with a life-threatening indication of RRT (defined as intractable hyperkalemia, acidosis, uremic symptoms) at enrollment,
  * RRT before recruitment,
  * known prehospitalization advanced chronic kidney disease (defined by an estimated GFR <30 mL/min/1.73 m2 or chronic RRT),
  * use of extracorporeal membrane oxygenation (ECMO),
  * diagnosis of hepatic cirrhosis or other condition with portal hypertension
  * Or postrenal causes of AKI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
assesment of KFR using the KDIGO AKI staging improvement | 1 week
  stage1:serum creatinine increase 1,5 - 2 folds serum creatinine increase 2 - 3 folds serum creatinine increase more than 3 folds

SECONDARY OUTCOMES:
VEXUS score | 48 hours
  grade 1 : no congestion grade 2:mild congestion grade 3 moderate congestion grade 4 : severe congestion

CONTACTS AND LOCATIONS:
Overall Officials: asmaa AS Behairy, master, Principal Investigator — Benha University
Locations (1):
- Asmaa Shahat Mohamedy Behairy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No